CLINICAL TRIAL: NCT02329769
Title: A Phase II, Open Label, Extension Study to Assess the Effect of PRO044 in Patients With Duchenne Muscular Dystrophy
Brief Title: Open Label, Extension Study of PRO044 in Duchenne Muscular Dystrophy (DMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO044-CLIN-02
Record Dates: First submitted 2014-12-22; First posted 2015-01-01 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy; DMD; BioMarin; PRO044
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRO044 SC 6 mg/kg (Experimental): Weekly subcutaneous (SC) dosing with 6 mg/kg
  Interventions: Drug: PRO044 SC 6 mg/kg
- PRO044 IV 6 mg/kg (Experimental): Weekly intravenous (IV) dosing with 6 mg/kg
  Interventions: Drug: PRO044 IV 6 mg/kg
- PRO044 SC 9 mg/kg (Experimental): Weekly intravenous (IV) dosing with 9 mg/kg
  Interventions: Drug: PRO044 IV 9 mg/kg

INTERVENTIONS:
Drug: PRO044 SC 6 mg/kg
  Arms: PRO044 SC 6 mg/kg
Drug: PRO044 IV 6 mg/kg
  Arms: PRO044 IV 6 mg/kg
Drug: PRO044 IV 9 mg/kg
  Arms: PRO044 SC 9 mg/kg

SUMMARY:
The purpose of this study is to see whether PRO044 is safe and effective to use as medication for Duchenne Muscular Dystrophy (DMD) patients with a mutation around location 44 in the DNA for the dystrophin protein.

DETAILED DESCRIPTION:
A Phase II, open-label, extesion study. Following a Screening period of up to one month, subjects previously treated with PRO044, and eligible for enrolment in PRO044-CLIN-02, will be allocated to one of three groups to receive either 6 mg/kg or 9 mg/kg PRO044 weekly by IV infusion or 6 mg/kg weekly by SC injection for 48 weeks.

Safety and tolerability, pharmacokinetics (PK), pharmacodynamic (PD) and efficacy assessments will be conducted at regular intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects previously treated with PRO044.
2. Continued use of glucocorticoids for a minimum of 60 days prior to study entry with a reasonable expectation that the subject will remain on steroids for the duration of the study. Changes to the dose regimen or cessation of glucocorticoids will be at the discretion of the Principle Investigator (PI) in consultation with the subject/parent and the Medical Monitor. If the subject is not on steroids, involvement in the study needs to be discussed with the medical monitor

Exclusion Criteria:

1. Current, or history of, liver or renal disease.
2. Acute illness within 4 weeks prior to the first dose of PRO044 (Week 1) which may interfere with the measurements.
3. Severe cardiac myopathy which in the opinion of the Investigator prohibits participation in this study
4. Need for daytime mechanical ventilation.
5. Screening aPTT above the upper limit of normal (ULN).
6. Screening platelet count below the lower limit of normal (LLN).
7. Use of anticoagulants, antithrombotics or antiplatelet agents.
8. Use of any investigational product within 6 months prior to the start of Screening for the study.
9. Current or history of drug and/or alcohol abuse.

Ages: 9 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of PRO044 (composite of several measures) | After 48 weeks of treatment
  Efficacy parameters:
  Muscle Function
  * 6 Minute Walk Distance (6MWD)
  * North Star Ambulatory Assessment
  * Timed tests (10-meter walk/run, rising from floor, stair climb)
  * DMD Functional Outcomes Questionnaire (DMD-FOS) -for ambulant subjects only
  * Egen Klassification - for non-ambulant subjects.
  Muscle strength
  * Pulmonary Function (Spirometry)
  * Handheld myometry.
  Exploratory:
  * Performance Upper Limb (PUL).
  * Patient Reported Outcome measure (PROM).
Safety and tolerability of PRO044 (treatement emergent adverse events) | After 48 weeks of treatment
  Number of subjects with 1 or more treatement emergent adverse events following SC or IV PRO044 dosing

SECONDARY OUTCOMES:
Assess the pharmacokinetics of PRO044 (composite of several measures) | After 48 weeks of treatment
  Pharmacokinetic parameters:
  * t ½
  * AUC: 0-24h, 0-∞ (where applicable)
  * Cmax
  * tmax
  * CL (for IV subjects) or CL/F (for SC subjects)
  * PRO044 concentrations in muscle tissue.

CONTACTS AND LOCATIONS:
Locations (5):
- UZ Leuven, Leuven, Belgium
- Italy (2):
  - S.Anna Hospital, Ferrara
  - Policlinico Universitario Agostino Gemelli, Roma
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Drottning Silvias Barn- ochungdomssjukhus, Gothenburg, Sweden